CLINICAL TRIAL: NCT03094052
Title: An Open Label Study to Characterize the Incidence and Severity of Diarrhea in Patients With HER2+ Breast Cancer Treated With Neratinib With or Without Trastuzumab
Brief Title: Incidence and Severity of Diarrhea in Patients With HER2 Positive Breast Cancer Treated With Trastuzumab and Neratinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Puma Biotechnology, Inc. (Industry)
Responsible Party: Principal Investigator, Jo Chien, Associate Clinical Professor of Medicine, University of California, San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 167514; NCI-2017-01443 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2017-03-14; First posted 2017-03-29 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: HER2-positive Breast Cancer; Breast Adenocarcinoma; Stage II Breast Cancer AJCC v6 and v7; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
Keywords: Neratinib; Trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib; Trastuzumab; Loperamide; crofelemer; atropine sulfate-diphenoxylate hydrochloride drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adjuvant Neratinib, Crofelemer, Loperamide (Experimental): Participants will receive 240mg neratinib to be taken continuously in 21-day cycles once a day for up to 55 weeks on study with no rest between cycles unless related to toxicity. Participants will receive Neratinib and may also be prescribed standard of care maintenance adjuvant trastuzumab (duration of maintenance trastuzumab is at the discretion of the treating physician), for up to 55 weeks. If applicable, after the completion of trastuzumab maintenance therapy (determined by treating physician), neratinib may continue as monotherapy to complete a maximum of 55 weeks. Participants will also receive 125mg of prophylactic Crofelemer and 4 mg of prophylactic loperamide as needed in the first 2 cycles.
  Interventions: Drug: Neratinib; Biological: Trastuzumab; Drug: Loperamide; Drug: Crofelemer; Drug: Diphenoxylate/Atropine
- Adjuvant Neratinib, Loperamide (Experimental): Participants will receive 120 mg of neratinib on days 1-7 with subsequent increase in dose by 40 mg every 7 days until the full dose of 240 mg a day is reached within the first cycle (up to 240mg) to be taken continuously in 21-day cycles once a day for up to 55 weeks on study with no rest between cycles unless related to toxicity. Participants will receive Neratinib and may also be prescribed standard of care maintenance adjuvant trastuzumab (duration of maintenance trastuzumab is at the discretion of the treating physician), for up to 55 weeks. If applicable, after the completion of trastuzumab maintenance therapy (determined by treating physician), neratinib may continue as monotherapy to complete a maximum of 55 weeks. Participants will also receive 4 mg of prophylactic loperamide to be taken as needed.
  Interventions: Drug: Neratinib; Biological: Trastuzumab; Drug: Loperamide

INTERVENTIONS:
Drug: Neratinib — Given orally (PO)
  Other Names: Nerlynx
Biological: Trastuzumab — Given Intravenously (IV)
  Other Names: Herceptin; HER2 Monoclonal Antibody
Drug: Loperamide — Given PO
  Other Names: Imodium
Drug: Crofelemer — Given PO
  Other Names: Mytesi
  Arms: Adjuvant Neratinib, Crofelemer, Loperamide
Drug: Diphenoxylate/Atropine — Allowed for participants experiencing refractory diarrhea
  Other Names: Lomotil
  Arms: Adjuvant Neratinib, Crofelemer, Loperamide

SUMMARY:
This phase II trial studies the incidence and severity of diarrhea in patients with stage II-IIIC HER2 Positive breast cancer treated with trastuzumab and neratinib. Trastuzumab is a form of targeted therapy because it attaches itself to specific molecules (receptors) on the surface of cancer cells, known as HER2 receptors. When trastuzumab attaches to HER2 receptors, the signals that tell the cells to grow are blocked and the cancer cell may be marked for destruction by the body's immune system. Neratinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving trastuzumab and neratinib may work better in treating patients with stage II-IIIC HER2 positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the incidence and severity of diarrhea in patients with early stage breast cancer receiving adjuvant neratinib with or without trastuzumab in the setting of anti-diarrheal strategies.

SECONDARY OBJECTIVES:

I. To evaluate the incidence of grade 3 or higher diarrhea using the dose-escalation strategy and anti-diarrhea medications as needed (prn) in patients who received prior trastuzumab emtansine (T-DM1).

II. To assess neratinib adherence, holds, delays, and early discontinuation throughout the course of study therapy which includes patients receiving neratinib for > 1 year.

III. To assess overall toxicity including constipation and cardiac toxicity with concomitant neratinib and trastuzumab.

OUTLINE: This is a dose-escalation study of neratinib. Patients receive one of the following treatment regimen:

NERATINIB MONOTHERAPY: Patients receive neratinib orally (PO) once daily (QD) on days 1-21. Cycles repeats every 21 days for up to 55 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive loperamide and/or diphenoxylate hydrochloride/atropine sulfate as needed per physician discretion for symptom management.

NERATINIB AND TRASTUZUMAB: Patients receive neratinib PO QD on days 1-21. Patients also receive trastuzumab maintenance therapy as determined by treating physician. Treatment repeats every 21 days for up to 55 weeks in the absence of disease progression or unacceptable toxicity. After completion of trastuzumab treatment, patients may continue on neratinib monotherapy for the remainder of the 55 weeks. Patients may receive loperamide and/or diphenoxylate hydrochloride/atropine sulfate as needed per physician discretion for symptom management.

After completion of studies treatment, patients are followed up for 28 days.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age >= 18 years
* Histologically confirmed clinical or pathological stage 2 through stage 3c primary adenocarcinoma of the breast
* Documented human epidermal growth factor receptor 2 (HER2) overexpression or gene-amplified tumor by a validated approved method
* Patients can have hormone receptor (HR)+ or HR-negative disease
* Concurrent adjuvant endocrine therapy and bone-modifying agents is allowed
* Patients can be premenopausal or postmenopausal
* Completion of neoadjuvant or adjuvant chemotherapy
* Completion of adjuvant locoregional radiation, if indicated, is required prior to starting study treatment
* Histologically confirmed clinical or pathological stage 2 through stage 3c primary adenocarcinoma of the breast
* Documented HER2 overexpression or gene-amplified tumor by a validated approved method
* Patients can have hormone receptor (HR)+ or HR-negative disease
* Concurrent adjuvant endocrine therapy and bone-modifying agents is allowed
* Patients can be premenopausal or postmenopausal
* Completion of neoadjuvant or adjuvant chemotherapy
* Completion of adjuvant locoregional radiation, if indicated, is required prior to starting study treatment
* At the time of study enrollment, patients can still be receiving adjuvant trastuzumab monotherapy or be within 2 years of completing adjuvant trastuzumab +/- pertuzumab maintenance, or adjuvant T-DM1.

  * Patients who are within 2 years of completing trastuzumab +/- pertuzumab or T-DM1 will receive neratinib monotherapy (and not neratinib + trastuzumab)
  * Adjuvant T-DM1 is the standard of care for patients who have residual disease after neoadjuvant chemotherapy. Patients with residual disease after neoadjuvant chemotherapy should receive T-DM1 before enrolling on the study. If not, the option of T-DM1 should be discussed with the patient
* Clinically no evidence of metastatic disease at the time of study entry. Patients with fully resected locoregional recurrence with no evidence of disease are eligible
* Left ventricular ejection fraction (LVEF) >= 50% measured by multiple-gated acquisition scan (MUGA) or echocardiogram (ECHO)
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 1
* Negative beta-human chorionic gonadotropin (hCG) pregnancy test for premenopausal women of reproductive capacity (those who are biologically capable of having children) and for women less than 12 months after menopause; (women are considered postmenopausal if they are >= 12 months without menses, in the absence of endocrine or anti-endocrine therapies)
* Trastuzumab can cause embryo-fetal harm when administered during pregnancy and the effects of neratinib on the developing human fetus are unknown. Women of child-bearing potential must agree and commit to use of a highly effective double-barrier method of contraception (e.g., a combination of male condom with an intravaginal device such as the cervical cap, diaphragm, or vaginal sponge with spermicide) or a non-hormonal method, from the signing of informed consent until 28 days after the last dose of neratinib and 7 months after the last dose of trastuzumab, or consent to total sexual abstinence (abstinence must occur from randomization and continue for 28 days after the last dose of neratinib and 7 months after the last dose of trastuzumab). Men without confirmed vasectomy must agree and commit to use a barrier method of contraception while on treatment and for 3 months after the last dose of investigational products, or consent to total sexual abstinence (abstinence must occur from randomization and continue for 3 months after the last dose of study medication)
* Recovery (i.e., to grade 1 or baseline) from all clinically significant adverse event (AE)s related to prior therapies (excluding alopecia, neuropathy, and nail changes)
* Provide written, informed consent to participate in the study and follow the study procedures

EXCLUSION CRITERIA:

* Clinical or radiologic evidence of metastatic disease prior to or at the time of study entry. Locoregional recurrent disease that is resected is allowed
* Currently receiving chemotherapy, radiation therapy, investigational immunotherapy, or investigational biotherapy for breast cancer
* Major surgery (including breast surgery) within < 30 days of starting treatment or received chemotherapy, investigational agents, or other cancer therapy < 14 days prior to the initiation of investigational products (except adjuvant endocrine therapy)
* Active uncontrolled cardiac disease, including cardiomyopathy, congestive heart failure (New York Heart Association functional classification of >= 2; including individuals who currently use digitalis, beta-blockers, or calcium channel blockers specifically for congestive heart failure), unstable angina, myocardial infarction within 12 months of enrollment, or ventricular arrhythmia
* Corrected QT (QTc) interval > 0.450 seconds (males) or > 0.470 seconds (females), or known history of QTc prolongation or Torsade de Pointes (TdP)
* Absolute neutrophil count (ANC) =< 1,000/microliter (uL)
* Platelets =< 100,000/uL
* Hemoglobin =< 9 g/dL
* Serum creatinine >= 1.5 x upper limit of normal (ULN) OR calculated creatinine clearance =< 30 mL/min for patients with creatinine levels > 1.5 x institutional ULN

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin >= 1.5 x ULN OR direct bilirubin >= ULN for patients with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase ([SGOT)) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase (SGPT)) >= 2.5 x ULN
* Second malignancy for which the patient will be receiving active treatment during the time of study participation.
* Currently pregnant or breast-feeding
* Significant chronic gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or grade >= 2 National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v.4.0) diarrhea of any etiology at baseline)
* Clinically active infection with hepatitis B or hepatitis C virus
* Evidence of significant medical illness, abnormal laboratory finding, or psychiatric illness/social situations that could, in the investigator's judgment, make the patient inappropriate for this study
* Known hypersensitivity to any component of the investigational products
* Unable or unwilling to swallow tablets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Chien, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Slamon DJ, Clark GM, Wong SG, Levin WJ, Ullrich A, McGuire WL. Human breast cancer: correlation of relapse and survival with amplification of the HER-2/neu oncogene. Science. 1987 Jan 9;235(4785):177-82. doi: 10.1126/science.3798106.
- [Background] Perez EA, Romond EH, Suman VJ, Jeong JH, Sledge G, Geyer CE Jr, Martino S, Rastogi P, Gralow J, Swain SM, Winer EP, Colon-Otero G, Davidson NE, Mamounas E, Zujewski JA, Wolmark N. Trastuzumab plus adjuvant chemotherapy for human epidermal growth factor receptor 2-positive breast cancer: planned joint analysis of overall survival from NSABP B-31 and NCCTG N9831. J Clin Oncol. 2014 Nov 20;32(33):3744-52. doi: 10.1200/JCO.2014.55.5730. Epub 2014 Oct 20. PMID 25332249
- [Background] Chan A, Delaloge S, Holmes FA, Moy B, Iwata H, Harvey VJ, Robert NJ, Silovski T, Gokmen E, von Minckwitz G, Ejlertsen B, Chia SKL, Mansi J, Barrios CH, Gnant M, Buyse M, Gore I, Smith J 2nd, Harker G, Masuda N, Petrakova K, Zotano AG, Iannotti N, Rodriguez G, Tassone P, Wong A, Bryce R, Ye Y, Yao B, Martin M; ExteNET Study Group. Neratinib after trastuzumab-based adjuvant therapy in patients with HER2-positive breast cancer (ExteNET): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2016 Mar;17(3):367-377. doi: 10.1016/S1470-2045(15)00551-3. Epub 2016 Feb 10. PMID 26874901
- [Background] Rabindran SK, Discafani CM, Rosfjord EC, Baxter M, Floyd MB, Golas J, Hallett WA, Johnson BD, Nilakantan R, Overbeek E, Reich MF, Shen R, Shi X, Tsou HR, Wang YF, Wissner A. Antitumor activity of HKI-272, an orally active, irreversible inhibitor of the HER-2 tyrosine kinase. Cancer Res. 2004 Jun 1;64(11):3958-65. doi: 10.1158/0008-5472.CAN-03-2868. PMID 15173008
- [Background] Burstein HJ, Sun Y, Dirix LY, Jiang Z, Paridaens R, Tan AR, Awada A, Ranade A, Jiao S, Schwartz G, Abbas R, Powell C, Turnbull K, Vermette J, Zacharchuk C, Badwe R. Neratinib, an irreversible ErbB receptor tyrosine kinase inhibitor, in patients with advanced ErbB2-positive breast cancer. J Clin Oncol. 2010 Mar 10;28(8):1301-7. doi: 10.1200/JCO.2009.25.8707. Epub 2010 Feb 8. PMID 20142587
- [Background] Martin M, Bonneterre J, Geyer CE Jr, Ito Y, Ro J, Lang I, Kim SB, Germa C, Vermette J, Wang K, Wang K, Awada A. A phase two randomised trial of neratinib monotherapy versus lapatinib plus capecitabine combination therapy in patients with HER2+ advanced breast cancer. Eur J Cancer. 2013 Dec;49(18):3763-72. doi: 10.1016/j.ejca.2013.07.142. Epub 2013 Aug 15. PMID 23953056
- [Background] Castro JG, Chin-Beckford N. Crofelemer for the symptomatic relief of non-infectious diarrhea in adult patients with HIV/AIDS on anti-retroviral therapy. Expert Rev Clin Pharmacol. 2015;8(6):683-90. doi: 10.1586/17512433.2015.1082424. Epub 2015 Aug 27. PMID 26517110
- [Background] Tradtrantip L, Namkung W, Verkman AS. Crofelemer, an antisecretory antidiarrheal proanthocyanidin oligomer extracted from Croton lechleri, targets two distinct intestinal chloride channels. Mol Pharmacol. 2010 Jan;77(1):69-78. doi: 10.1124/mol.109.061051. Epub 2009 Oct 6. PMID 19808995
- [Background] Crutchley RD, Miller J, Garey KW. Crofelemer, a novel agent for treatment of secretory diarrhea. Ann Pharmacother. 2010 May;44(5):878-84. doi: 10.1345/aph.1M658. Epub 2010 Apr 13. PMID 20388859
- [Background] Macarthur RD, Hawkins TN, Brown SJ, Lamarca A, Clay PG, Barrett AC, Bortey E, Paterson C, Golden PL, Forbes WP. Efficacy and safety of crofelemer for noninfectious diarrhea in HIV-seropositive individuals (ADVENT trial): a randomized, double-blind, placebo-controlled, two-stage study. HIV Clin Trials. 2013 Nov-Dec;14(6):261-73. doi: 10.1310/hct1406-261. PMID 24334179

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 0 | 1 | 1
  40-49 years old | 6 | 0 | 6
  50-59 years old | 0 | 3 | 3
  60-69 years old | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11
Hormone receptor positive (HR+) [Number; unit: participants] — Breast cancer cells that have receptors for either estrogen or progesterone are considered hormone receptor-positive (HR+).
  participants | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 3 or Greater Diarrhea
Description: Percentage of participants with clinically assessed grade 3 or greater diarrhea reported within the first 2 cycles (each cycle is 21 days) of neratinib while using anti-diarrheal strategies. Reports of diarrhea will be graded according to NCI CTCAE version 4.0.
Time Frame: Up to 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
percentage of participants | 29 | 50

2. Primary Outcome: Percentage of Participants Who Did Not Require Loperamide During Multiple Cycles of Treatment
Description: Percentage of participants who did not require loperamide during cancer treatment for at least 5 cycles will be reported.
Time Frame: Up to 55 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
percentage of participants | 71 | 50

3. Primary Outcome: Percentage of Participants Who Discontinued Anti-diarrheal Medications for Multiple Cycles of Treatment
Description: The percentage of participants who discontinued all anti-diarrheal medications during cancer treatment for at least 5 cycles will be reported.
Time Frame: Up to 55 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
percentage of participants | 43 | 25

4. Primary Outcome: Percentage of Participants With Treatment-related Adverse Events
Description: Percentage of participants with reported serious adverse events and adverse events of interest of any grade that have been determined to be related to the anti-diarrhea treatment will be reported by worst grade and associated toxicity.
Time Frame: Up to 55 weeks
Population: All participants experienced only Grade 1, Constipation related to anti-diarrhea medication. No other treatment-related adverse events were reported.
Measure: Number; unit: percentage of participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
percentage of participants | 100 | 100

5. Primary Outcome: Number of Participants With Neratinib Dose Holds
Description: The number of participants who experienced a dose hold of neratinib during the course of study therapy will be reported
Time Frame: Up to 55 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
Participants | 0 | 0

6. Primary Outcome: Number of Participants Who Discontinued Neratinib Early
Description: The number of participants who discontinued neratinib earlier than expected during the course of study therapy will be reported
Time Frame: Up to 55 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
Participants | 1 | 0

7. Primary Outcome: Number of Participants With Neratinib Dose-reductions
Description: The number of participants whose dose was reduced at any time during the course of therapy will be reported
Time Frame: Up to 55 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
Number analyzed (Participants) | 7 | 4
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Up to 55 weeks
Arm/Group | Adjuvant Neratinib, Crofelemer, Loperamide | Adjuvant Neratinib, Loperamide
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 7/7 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjuvant Neratinib, Crofelemer, Loperamide (N=7) | Adjuvant Neratinib, Loperamide (N=4)
Diarrhea (Gastrointestinal disorders) | 7 (163) | 4 (56)
Constipation (Gastrointestinal disorders) | 7 (68) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 4 (13) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 1 (2)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (6) | 2 (2)
Fever (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (2) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 3 (3) | 0 (0)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (2) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study closed to enrollment earlier than expected due to a change in pharmaceutical sponsor priorities and treatment landscape.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03094052/Prot_SAP_000.pdf